CLINICAL TRIAL: NCT00761891
Title: Validation of an Ex Vivo Cyclooxygenase-1 Catalytic Assay in Humans
Brief Title: Validation of an Assay to Measure Cyclooxygenase-1 Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, John Oates, Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 061190
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: aspirin; cyclooxygenase-1; aspirin resistance; aspirin nonresponse; platelet; Normal volunteers
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chewable aspirin (Experimental): 81 mg daily for 2 weeks
  Interventions: Other: Chewable aspirin

INTERVENTIONS:
Other: Chewable aspirin — chewable aspirin 81mg daily for 2 weeks
  Other Names: acetylsalicylic acid

SUMMARY:
The purpose of this study is to obtain a reference range for a newly developed assay of ex vivo platelet COX-1 activity in normal volunteers taking a routine clinical dose of aspirin.

DETAILED DESCRIPTION:
Aspirin has been shown to reduce cardiovascular events in at-risk individuals, but some aspirin-treated patients fail to exhibit expected changes in bleeding time and platelet aggregation. Recent evidence has correlated aspirin "non-response" to poor cardiovascular outcomes.

In order to study the mechanisms of aspirin resistance, an assay is needed to measure the catalytic activity of platelet cyclooxygenase (which should be inhibited by aspirin). A common assay in general use is the measurement of thromboxane B2 production in clotting whole blood. This measure, however, is influenced by genetic and environmental variations in the glass-activated coagulation pathway, albumin binding capacity, platelet activation pathways, arachidonic acid pools, and phospholipase activity.

Our laboratory has developed a direct assay of platelet cyclooxygenase (COX-1) activity that is not influenced by these variations. This study will generate a reference range in normal volunteers taking a routine clinical dose of aspirin (81mg daily) for this assay.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker
* No chronic medical illness
* No chronic medications

Exclusion Criteria:

* Aspirin/NSAID use in preceding 14 days
* History of chronic NSAID use
* Currently taking NSAIDs, opioid analgesics, corticosteroids, or anticoagulants
* History of coronary artery disease, myocardial infarction, coronary artery bypass grafting, percutaneous angioplasty, diabetes mellitus, or stroke.
* History of hypertension
* Body mass index > 35
* History of gastric, duodenal, or esophageal ulcers or serious gastrointestinal bleed
* History of frequent headaches, pain syndrome, or other condition requiring frequent use of analgesics
* History of adverse reactions to aspirin
* Screening platelet count < 100,000/ul or > 500,000/ul
* Screening hematocrit < 35% or > 50%
* Weight less than 110 pounds
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-05; Primary Completion 2008-05 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Oates, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chewable Aspirin
Started | 64
Completed | 54
Not Completed | 10
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Arm/Group | Chewable Aspirin
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 33.5 [18 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 38
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: A Reference Range in Normal Volunteers Taking a Routine Clinical Dose of Aspirin (81mg Daily) for 2 Weeks
Description: Determine the level of Thromboxane B2 at which patients with a result above are not fully inhibited, and patients with a TxB2 level below are fully inhibited.
  The reference range is the level of serum thromboxane at which participants below have fully inhibited COX-1 and participants above do not have fully inhibited COX-1 activity
Time Frame: 2 weeks
Measure: Number (75% Confidence Interval); unit: ng/ml
Arm/Group | Chewable Aspirin
Number analyzed (Participants) | 54
ng/ml | 13 [4.988 to 13]

2. Secondary Outcome: Serum Thromboxane
Description: SerumTxB2: They are formed from the prostaglandin endoperoxides and cause platelet aggregation, contraction of arteries, and other biological effects.
Time Frame: Baseline and at 2 weeks
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- Chewable Aspirin: 81mg aspirin daily for 2 weeks
Arm/Group | Chewable Aspirin
Number analyzed (Participants) | 54
ng/ml
  baseline | 284.2 (11.53)
  2weeks | 9.542 (0.92)

ADVERSE EVENTS:
Groups:
- Enteric-coated Aspirin: 81 mg daily for 2 weeks
  Enteric-coated aspirin: enteric-coated aspirin 81mg daily for 2 weeks
Arm/Group | Enteric-coated Aspirin
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No